CLINICAL TRIAL: NCT00061022
Title: SAINT (Stroke - Acute Ischemic - NXY Treatment) A Double Blind, Randomized, Placebo Controlled, Parallel Group, Multicenter, Phase IIb/III Study to Assess the Efficacy and Safety of Intravenous NXY-059 in Acute Ischemic Stroke
Brief Title: Safety and Effectiveness of NXY-059 for the Treatment of Patients Who Have Suffered From a Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: SA-NXY-0007; 007; SAINT 2
Record Dates: First submitted 2003-05-20; First posted 2003-05-21 (Estimated); Last update posted 2010-11-15 (Estimated); Status verified 2010-11

CONDITIONS: Cerebral Stroke; Stroke, Acute; Cerebrovascular Stroke; Ischemic Attack, Transient
Keywords: Stroke; cerebral vascular accident; CVA; Ischemia; Hemorrhage; TIA; Transient Ischemic Attack; Brain Attack; Cataplexy
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Ischemia; Hemorrhage; Cataplexy | interventions — disufenton sodium

INTERVENTIONS:
Drug: NXY-059

SUMMARY:
This study will determine if NXY-059 will improve recovery from an acute stroke. The study is designed to look at both overall recovery and recovery of motor function, for example muscle strengthen and coordination.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Acute ischemic stroke with limb weakness
* Onset of symptoms within 6 hours
* Full functional independence prior to the present stroke

Exclusion Criteria:

* Unconsciousness
* Subjects who are unlikely to complete the infusion of investigational product and/or are unlikely to undergo active medical management during that period due to a severe clinical condition.
* Severe illness with life expectancy less than 6 months.
* Known severe kidney disorder.
* Current known alcohol or illicit drug abuse or dependence.
* Pregnant or breast-feeding.
* Treatment with acetazolamide and methotrexate is not permitted during the infusion
* Participation in a previous clinical study within 30 days.
* Meets all other exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200
Dates: Start 2003-05; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Global disability on modified Rankin scale at 90 days.

SECONDARY OUTCOMES:
NIH stroke scale
Barthel Index
Stroke Impact Scale
EQ-5D all at 90 days
Safety outcomes

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca NXY-059 Medical Science Director, MD, Study Director — AstraZeneca
Locations (256):
- United States (98):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Fort Smith, Arkansas
  - Research Site, Arcadia, California
  - Research Site, Concord, California
  - Research Site, Englewood, California
  - Research Site, La Jolla, California
  - Research Site, La Mesa, California
  - Research Site, Los Angeles, California
  - Research Site, Oceanside, California
  - Research Site, Palo Alto, California
  - Research Site, Poway, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Englewood, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Fairfield, Connecticut
  - Research Site, Delray Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Lane Panama City, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Naples, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Weston, Florida
  - Research Site, Decatur, Georgia
  - Research Site, Lithonia, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Des Plaines, Illinois
  - Research Site, Elk Grove Village, Illinois
  - Research Site, Maywood, Illinois
  - Research Site, Oak Park, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Cedar Rapids, Iowa
  - Research Site, Des Moines, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, Marrero, Louisiana
  - Research Site, South Weymouth, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, East Lansing, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Golden Valley, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Reno, Nevada
  - Research Site, Edison, New Jersey
  - Research Site, Long Branch, New Jersey
  - Research Site, Lumberton, New Jersey
  - Research Site, Morristown, New Jersey
  - Research Site, Neptune City, New Jersey
  - Research Site, Red Bank, New Jersey
  - Research Site, Ridgewood, New Jersey
  - Research Site, Summit, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Trenton, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Flushing, New York
  - Research Site, New Hyde, New York
  - Research Site, Rochester, New York
  - Research Site, Schenectady, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Tualatin, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Beaufort, South Carolina
  - Research Site, Bristol, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Virginia Beach, Virginia
  - Research Site, Olympia, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Marshfield, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (6):
  - Research Site, Boulogne Sur Mer
  - Research Site, Buenos Aires
  - Research Site, Capital Federal
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mar del Plata
- Australia (7):
  - Research Site, Bedford Park
  - Research Site, Box Hill
  - Research Site, Camperdown
  - Research Site, Gosford
  - Research Site, Heidelberg
  - Research Site, New Lambton
  - Research Site, Parkville
- Austria (5):
  - Research Site, Klosterneuburg
  - Research Site, Linz
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, Leuven
- Brazil (6):
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São Paulo
- Bulgaria (5):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Canada (21):
  - Research Site, Barrie
  - Research Site, Calgary
  - Research Site, Edmonton
  - Research Site, Greenfield Park
  - Research Site, Halifax
  - Research Site, Kitchener
  - Research Site, Lethbridge
  - Research Site, Lévis
  - Research Site, Mississauga
  - Research Site, Montreal
  - Research Site, Ottawa
  - Research Site, Penticton
  - Research Site, Québec
  - Research Site, Saint John
  - Research Site, Saskatoon
  - Research Site, Thunder Bay
  - Research Site, Toronto
  - Research Site, Trois-Rivières
  - Research Site, Vancouver
  - Research Site, Victoriaville
  - Research Site, Windsor
- Research Site, Santiago, Chile
- China (3):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Shanghai
- Czechia (6):
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Pardubice
  - Research Site, Pelhřimov
  - Research Site, Prague
- France (13):
  - Research Site, Belfort
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Bourg-en-Bresse
  - Research Site, Créteil
  - Research Site, Le Chesnay
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Montbéliard
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Perpignan
  - Research Site, Toulouse
- Germany (6):
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Minden
  - Research Site, Wiesbaden
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Chai Wan
  - Research Site, Hong Kong
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kistarcsa
- Israel (11):
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
  - Research Site, Zrifin
- Mexico (6):
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Guadalajara
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Luis Potosí City
  - Research Site, Zapopan, Jalisco
- Research Site, Grafton, New Zealand
- Philippines (3):
  - Research Site, Manila
  - Research Site, Pasay
  - Research Site, Quezon City
- Poland (12):
  - Research Site, Częstochowa
  - Research Site, Gdansk
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Opole
  - Research Site, Siedlce
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Zabrze
- Portugal (5):
  - Research Site, Amadora
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Setúbal
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Slovakia (4):
  - Research Site, Lovoca
  - Research Site, Martin
  - Research Site, Nitra
  - Research Site, Ziliha
- South Africa (4):
  - Research Site, Cape Town
  - Research Site, George
  - Research Site, Morningside
  - Research Site, Somerset West
- South Korea (2):
  - Research Site, Anyang
  - Research Site, Seoul
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Santiago(A Coruña)
- Switzerland (6):
  - Research Site, Aarau
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Lausanne
  - Research Site, Sankt Gallen
  - Research Site, Zurich
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan Hsien
- United Kingdom (3):
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Newcastle upon Tyne

REFERENCES:
- [Derived] Shuaib A, Lees KR, Lyden P, Grotta J, Davalos A, Davis SM, Diener HC, Ashwood T, Wasiewski WW, Emeribe U; SAINT II Trial Investigators. NXY-059 for the treatment of acute ischemic stroke. N Engl J Med. 2007 Aug 9;357(6):562-71. doi: 10.1056/NEJMoa070240. PMID 17687131